CLINICAL TRIAL: NCT00000777
Title: Active Immunization of HIV-1 Infected, Pregnant Women With CD4 Lymphocyte Counts >= 400/mm3: A Phase I Study of Safety and Immunogenicity of VaxSyn Recombinant gp160 (NOTE: Some Patients Receive Placebo)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Model: Parallel | Purpose: Treatment
Other Study IDs: ACTG 234; VEU 102; 11211 (Registry Identifier: DAIDS ES Registry Number)
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2021-10-28 (Actual); Status verified 2021-10

CONDITIONS: HIV Infections; Pregnancy; HIV Seronegativity
Keywords: Vaccines, Synthetic; Pregnancy; Pregnancy Complications, Infectious; HIV Envelope Protein gp160; AIDS Vaccines; HIV Preventive Vaccine; HIV Therapeutic Vaccine
MeSH Terms: conditions — HIV Infections; Pregnancy Complications, Infectious | interventions — VaxSyn HIV-1 (gp160) vaccine

INTERVENTIONS:
Biological: gp160 Vaccine (MicroGeneSys)

SUMMARY:
To evaluate the safety of gp160 vaccine (VaxSyn) in HIV-1 infected pregnant women with CD4 counts >= 400 cells/mm3. To evaluate the immunogenicity of this vaccine in pregnant women and the passive acquisition of vaccine-specific antibody in their infants.

Evidence suggests that an advanced stage of disease with high plasma viremia is associated with increased transmission of HIV-1 to the fetus. Slowing the progression of disease, reducing the titer of virus in plasma, and increasing the titer of epitope-specific antibody are potentially attainable goals through active immunization of the mother during pregnancy.

DETAILED DESCRIPTION:
Evidence suggests that an advanced stage of disease with high plasma viremia is associated with increased transmission of HIV-1 to the fetus. Slowing the progression of disease, reducing the titer of virus in plasma, and increasing the titer of epitope-specific antibody are potentially attainable goals through active immunization of the mother during pregnancy.

Pregnant women are randomized to receive an initial injection of VaxSyn or alum placebo between week 16 and week 24 of gestation, followed by monthly booster injections concluding at the end of pregnancy, for a total of five injections. Patients may have optional booster immunizations (vaccine or placebo) at 3, 6, 9, and 12 months after delivery. Mothers and infants are followed through 18 months after delivery.

ELIGIBILITY:
Inclusion Criteria

Concurrent Medication:

Allowed:

* AZT.
* Acyclovir.

Patients must have:

* HIV-1 infection.
* CD4 count >= 400 cells/mm3.
* No AIDS-defining illness or other systemic manifestations related to HIV (other than generalized lymphadenopathy).
* HIV p24 < 30 pg/ml.
* Proven pregnancy in the 16th to 24th week of gestation at study entry, with no special obstetrical risks.
* Concurrent AZT therapy is permitted.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms and conditions are excluded:

* Known hypersensitivity to a component of the vaccine.
* Evidence of fetal abnormality on ultrasound.
* Evidence of maternal risk factors including insulin-dependent diabetes, moderate to severe hypertension, repeated fetal wastage (> 3), Rh-sensitization or other blood group alloimmunization, severe renal disease, previous infants with malformations or other factors that obstetrically are judged to constitute a special risk of spontaneous abortion or premature birth.
* Active syphilis.
* Hepatitis B surface antigen positive.

Concurrent Medication:

Excluded:

* Antiretroviral or immunomodulating agent other than AZT during the pregnancy.

Prior Medication:

Excluded:

* Antiretroviral or immunomodulating agent other than AZT within 90 days prior to study entry.

Current use of illicit drugs or known chronic alcohol use.

Ages: 16 Years to 40 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 24
Dates: Study Completion 1998-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Sullivan JL, Study Chair; Lambert JS, Study Chair; Wright PF, Study Chair
Locations (2):
- United States (2):
  - Yale Univ Med School, New Haven, Connecticut
  - Vanderbilt Univ Hosp, Nashville, Tennessee